CLINICAL TRIAL: NCT07006142
Title: Effect of Prolonged Fasting Time on Gastric Residual Volume in Patients Taking GLP1 Receptor Agonists
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Krishnan Ramanujan, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: 23-013192
Record Dates: First submitted 2025-05-27; First posted 2025-06-05 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Upper Endoscopy; GLP1-R-related Disease
Keywords: GLP1 receptor agonists; upper endoscopy

STUDY DESIGN:
Intervention Model Description: This study has 3 arms, but two of them are historical cohorts (i.e. previous patients who have already been taken care of). One group will consist of patients who are not on GLP1 medications who underwent upper endoscopy, and another group will consist of patients who are on GLP1 medications who underwent upper endoscopy. The third group is the prospective group who are being enrolled and recruited - this group will consist of patients who are on GLP1 medications who abide by a modified fasting guideline consisting of a full-liquid diet 48 hours prior to procedure, clear liquid diet 24 hours prior to procedure, and no liquids or solids after midnight on the day of upper endoscopy.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Normal fasting guidelines and not taking GLP1-RAs (No Intervention): Patients who are not taking GLP1 RAs (Receptor Agonists) and who will abide by the normal fasting guidelines
- Normal fasting guidelines with GLP1-RAs (No Intervention): Patients who are taking GLP1 RAs (Receptor Agonists) for either diabetes or weight loss management who will abide by normal fasting guidelines
- Modified fasting guidelines with GLP1-RAs (Experimental): Patients who are prescribed and taking GLP1 RAs (Receptor Agonists) for either diabetes or weight loss management who follow the modified fasting guidelines. Modified fasting consists of a full-liquid diet 48 hours prior to the procedures, clear liquid diet 24 hours prior to their procedure, and nothing by mouth (NPO) after midnight on the day of their procedure.
  Interventions: Other: Modified Fasting Guidelines

INTERVENTIONS:
Other: Modified Fasting Guidelines — Patients will follow a full-liquid diet 48 hours prior to their procedure, clear liquid diet 24 hours prior to their procedure, and nothing by mouth (NPO) after midnight on the day of their procedure
  Arms: Modified fasting guidelines with GLP1-RAs

SUMMARY:
The aim of this study is to determine whether a modified fasting protocol can reduce the potential risk of aspiration for patients currently prescribed GLP1-RAs.

DETAILED DESCRIPTION:
The overall objective of this project is to identify a reasonable means by which patients on GLP1-RAs can be safely cared for in the perioperative period that can be agreed upon by all groups involved in perioperative patient care. This will be assessed in patients undergoing upper endoscopy specifically since assessment of gastric contents would be minimally invasive for this patient population receiving anesthetic care.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective upper endoscopy with gastroenterology team

Exclusion Criteria:

* Urgent or emergent procedure
* Inclusion of colonoscopy or antegrade small bowel enteroscopy in planned procedure
* Upper GI barium study performed in past 24 hours.
* Gastroparesis
* Achalasia
* Pancreatitis
* Use of outpatient pro-motility medications
* Patient refusal
* Inability for patient to provide own consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Gastric contents | Baseline
  Number of patients who were found to have gastric contents within the stomach during the upper endoscopy.

SECONDARY OUTCOMES:
Diagnosis of aspiration within 72 hours of procedure | From the time of upper endoscopy until 72 hours post-procedure.
  Whether or not a patient was diagnosed with aspiration will be determined via chart review for 72 hours after the completion of upper endoscopy. A note documenting aspiration or an ICD code associated with aspiration will indicate that this outcome occurred.
Aspiration pneumonitis diagnosis postoperatively | 72 hours after completion of upper endoscopy
  The number of patients who have a diagnosis of aspiration pneumonitis, as identified by the presence of ICD codes J69.0 or J69.8, postoperatively.
Postprocedural ICU admission | Immediately after upper endoscopy
  The number of patients who were admitted to the ICU immediately after upper endoscopy.

CONTACTS AND LOCATIONS:
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No